CLINICAL TRIAL: NCT00845234
Title: Establishing a Standard for Peri-operative ICD Patient Education: A Demonstration Project
Brief Title: Establishing a Standard for Peri-operative Implantable Cardioverter Defibrillator (ICD) Patient Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Aurora Denver Cardiology Associates (Unknown); Medtronic (Industry)
Responsible Party: Principal Investigator, Samuel F. Sears, Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00293-2008-0356-1
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Arrhythmia
Keywords: behavioral intervention; implantable cardioverter defibrillator; psychosocial education; anxiety; depression
MeSH Terms: conditions — Arrhythmias, Cardiac; Anxiety Disorders; Depression | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care Group (No Intervention): Received the current standard of care as operationally defined by the investigators- Q&A session + Video
- Intervention Group (Experimental): Intervention group- Patients will receive the brief educational CBT intervention + video and Q&A session
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Intervention consisted of a brief, educational CBT intervention and included the following domain areas: ICD knowledge and post-discharge care, understanding shock, stress management, family and relationships, device recall, and survivorship. The intervention was provided at baseline (0 weeks). Intervention was led by investigator and lasted 15 minutes in duration.
  Arms: Intervention Group

SUMMARY:
An implantable cardioverter defibrillator (ICD) administers a shock to terminate potentially life-threatening cardiac arrhythmias. The device saves lives, but presents psychological challenges for patients. At present, there is a paucity of brief interventions for ICD patients designed for administration in a clinic setting that considers issues of cost, time, and available resources. The present study examined the impact of a brief cognitive behavioral (CBT) educational intervention on primary endpoints of patient acceptance and quality of life and secondary endpoints of depression and anxiety. It was hypothesized that the intervention would result in significant improvements primary and secondary endpoints for participants in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* literate
* newly implanted with an implantable cardioverter defibrillator (ICD)

Exclusion Criteria:

* documented neurological sequelae associated with CVA or dementia
* documented cognitive impairment
* reported illiteracy
* previously implanted ICD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Score on measure assessing construct of quality of life | Up to 8 months after enrollment
  Quality of life will be obtained via participants scores from the Medical Outcomes Survey Short Form-12 (SF-12) measure of quality of life.

SECONDARY OUTCOMES:
Score on measure assessing depression | Up to 8 months after enrollment
  Depression will be assessed via participant's self-reported scores on the depression subscale of the Hospital Anxiety and Depression Scale (HADS).
score on measure assessing construct of patient acceptance of device | up to 8 months after enrollment
  The Florida Patient Acceptance Scale measures patient's self-reported acceptance of the implantable cardioverter defibrillator.
score on measure assessing anxiety | Up to 8 months after enrollment
  The Hospital Anxiety and Depression Scale is comprised of two subscales- anxiety and depression. It is a self-report measure that generates a score on the patient's current level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel F Sears, Ph.D., Principal Investigator — East Carolina University
Locations (3):
- United States (3):
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Aurora Denver Cardiology Associates, Lone Tree, Colorado
  - East Carolina Heart Institute, Greenville, North Carolina